CLINICAL TRIAL: NCT02820428
Title: Evaluation Comportementale Dans la Maladie de Parkinson. Normes Chez Des Sujets Sains
Brief Title: Evaluation of Behaviour in Parkinson's Disease. Normal Values in Healthy Subjects
Acronym: ECMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2009-A00103-54/3
Record Dates: First submitted 2016-05-25; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-05

CONDITIONS: Behaviour
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy participants (Other): Submission of the scale 'Evaluation of behaviour in Parkinson's Disease' to healthy subjects
  Interventions: Other: Healthy participants

INTERVENTIONS:
Other: Healthy participants — Semi-structured interview

SUMMARY:
Non-motor symptoms like mood fluctuations and behavioral disorders are frequent in Parkinson's disease. They may be induced by both the pathology and the dopaminergic treatment and must be considered in treatment policies.

Due to their specificity and the absence of an appropriate evaluation tool, behavioral disorders are rarely searched for.

Therefore, investigators developed a scale permitting qualitative and quantitative evaluation of behavior according to the severity of the disorders.

This study aims to define reference values for healthy individuals

DETAILED DESCRIPTION:
The application of the scale includes a semi-structured interview

The ECMP scale consists of 21 items, each of which may be assessed by use of a 5 point scale (not at all - light trouble - moderate trouble - important trouble - severe trouble)

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants without any neurologic disease
* Men and women from 25 to 75 years old
* French mother tong
* without cognitive troubles (MMS ≥ 24)

Exclusion Criteria:

* Subject under legal guardianship
* Pregnant woman or with childbearing potential without contraceptive device

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
ECMP score | 3 hours
  Semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Anna Castrioto, MD, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No